CLINICAL TRIAL: NCT03157986
Title: Effects of a Three Week Whole Body Vibration Training Versus Conventional Balance Training in Patients With Severe Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Whole-Body Vibration Training Versus Balance Training in Patients With Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Head physican (department of pneumology), Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WBVT Balance Study
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Balance; Whole Body Vibration Training; pulmonary rehabilitation; exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Body Vibration training (Active Comparator): Balance Training on a Vibration platform
  Interventions: Other: Balance Training on a vibration platform
- Conventional Balance training (Active Comparator): Balance Training on a Balance board
  Interventions: Other: Conventional Balance training

INTERVENTIONS:
Other: Balance Training on a vibration platform — n=24 patients with severe chronic obstructive pulmonary disease. Exercises will be performed on a side-alternating Vibration platform (Galileo) at frequencies between 15 to 26 Hertz.
  Arms: Whole Body Vibration training
Other: Conventional Balance training — n=24 patients with COPD, Exercises will be performed on a Balance pad
  Arms: Conventional Balance training

SUMMARY:
Aim of this study is to compare the effects of whole-body Vibration Training versus conventional Balance Training on Balance performance, gait quality and exercise capacity in patients with severe chronic obstructive pulmonary disease. Patients will be recruited during a 3-week inpatient pulmonary rehabilitation program and will be randomized into one of two intervention groups. On top of a standardized endurance and strength Training program (5 days per week) patients in both groups will perform an additional Balance Training (on 3 days per week). Patients in both Groups will perform the same 4 different Balance exercises (2x1 Minute each): dynamic squats with closed eyes, heel raise, semi-Tandem stance and single leg stance but on a different surface. The Vibration Training Group will perform the exercises on a side-alternating Vibration platform (Galileo) at frequencies between 15 to 26 Hertz and the control Group will perform exercises on instable objects like Balance pads. The degree of difficulty in both Groups will be individually adjusted and will be progressively increased, if possible.

ELIGIBILITY:
Inclusion Criteria:

* COPD stage III or IV according to the global initiative for chronic obstructive lung disease
* impaired exercise capacity (6 Minute walk distance of less than 70% of the reference value from Troosters et al.)

Exclusion Criteria:

* current acute exacerbation of COPD
* carbon dioxide pressure of more than 45 mmHg at rest
* any contraindication for vibration Training (e.g. acute deep vein thrombosis)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Change in Balance Performance during semi Tandem stance | measurement on Day 1 and 21
  patients stand still for 10 seconds with closed eyes on a force platform that measures absolute path length of the center of force.

SECONDARY OUTCOMES:
Change in muscle power during counter movement jump | measurement on Day 1 and 21
  patients jump on a force platform as high as possible. The Outcome is Watt per Kilogram Body weight
Change in performance of the 5-Repetition-Raise-Test | measurement on Day 1 and 21
  Patients try to perform 5 repetitions of standing up and sitting down from a chair with crossed arms on a force platform as quick as possible
Change in performance of the 1-Minute-Chair-Rise-Test | measurement on Day 1 and 21
  Patients try to perform as many repetitions as possible of standing up and sitting down from a chair with crossed arms on a force platform during 1 minute
Change in Peak muscle strength of the knee Extension muscles | measurement on Day 1 and 21
  isometric peak torque of the knee extensor muscles are measured in 90° knee angle
Change in Peak muscle strength of the knee Flexion muscles | measurement on Day 1 and 21
  isometric peak torque of the knee flexor muscles are measured in 90° knee angle
Change in 6-minute Walk Distance | measurement on Day 1 and 21
  patients are advised to walk as far as possible on a 30m track
Change in 4m Gait Speed Test | measurement on Day 1 and 21
  patients have to walk 4 meters at their usual Speed. Outcome is the average Speed during the 4m walk.
Change in step symmetry during 20m walking | measurement on Day 1 and 21
  Patients walk 20m while wearing the Mc Roberts move test device (triaxial accelerometer) which performs a gait analysis
Change in Hospital anxiety and Depression scale | measurement on Day 1 and 21
  the Hospital anxiety and Depression scale is a questionnaire that evaluates signs of anxiety or depression
Change in balance performance during Romberg stance | measurement on Day 1 and 21
  patients stand still for 10 seconds with closed eyes on a force platform that measures absolute path length of the center of force.
Change in Balance Performance during 1-leg stance | measurement on Day 1 and 21
  patients stand still for 10 seconds with closed eyes on a force platform that measures absolute path length of the center of force.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, MD, Principal Investigator — Schoen Klinik Berchtesgadener Land
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau am Königssee, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gloeckl R, Schneeberger T, Leitl D, Reinold T, Nell C, Jarosch I, Kenn K, Koczulla AR. Whole-body vibration training versus conventional balance training in patients with severe COPD-a randomized, controlled trial. Respir Res. 2021 May 4;22(1):138. doi: 10.1186/s12931-021-01688-x. PMID 33947416